CLINICAL TRIAL: NCT05741307
Title: Effect of a Self-hypnosis Smartphone Application on Attention Disorders and Anxiety in Children With Attention Deficit/Hyperactivity Disorder (ADHD)
Brief Title: Effect of a Self-hypnosis on Attention Disorders and Anxiety in Children With Attention Deficit/Hyperactivity Disorder
Acronym: HYPNAAX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: APHP220842; 2022-A01509-34 (Other: IDRCB Number)
Record Dates: First submitted 2022-11-03; First posted 2023-02-23 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Attention Deficit/Hyperactivity Disorder
Keywords: Attention Deficit/Hyperactivity Disorder; Anxiety; Hypnosis; Smartphone application; ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Anxiety Disorders | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients 2 (Experimental): Patient aged 7 to 12 with a diagnosis of ADHD made by a child psychiatrist or neuropediatrician and followed by the child psychiatry department - Reference Center for Language and Learning Disorders of the Necker Enfants Malades Hospital.
  These patients will use of the self-hypnosis application 6 weeks after inclusion : from T2 to T3.
  Interventions: Behavioral: Self-hypnosis application; Other: Questionnaires
- Patients 1 (Experimental): Patient aged 7 to 12 with a diagnosis of ADHD made by a child psychiatrist or neuropediatrician and followed by the child psychiatry department - Reference Center for Language and Learning Disorders of the Necker Enfants Malades Hospital.
  These patients will use of the self-hypnosis application at inclusion : from T0 (inclusion) to T1.
  Interventions: Behavioral: Self-hypnosis application; Other: Questionnaires

INTERVENTIONS:
Behavioral: Self-hypnosis application — The Hypnotidoo application offers screenless self-hypnosis sessions for 5-12 year olds. Each session lasts 6 to 8 minutes and focuses on one of the following themes: stress and anxiety, sleep, daily troubles and discomforts, hypersensitivity, hyperactivity and difficulty concentrating, self-confidence, difficult life events, anger. Each session begins with breathing and refocusing work, followed by self-hypnosis through stories and metaphors suitable for children.
  The application will be used by patients in the context of research for 6 weeks, 5 days out of 7 in parallel with the usual treatment.
  Other Names: Hypnotidoo application
Other: Questionnaires — Before and after (at T0, T1, T2 and T3) the 6-week period of use of the application and a wash-out period of 2 weeks (= usual treatment only), self- and hetero-questionnaires which constitute the gold standard for evaluating the symptoms of inattention and anxiety are proposed: Conners III, Child Behavior Checklist (CBCL) and Revised-Children's Manifest Anxiety Scale (R-CMAS).
  * T0: inclusion
  * T1: 6 weeks after T0 (inclusion)
  * T2: 2 weeks after T1
  * T3: 6 weeks after T2
  Other Names: Conners III, CBCL and R-CMAS

SUMMARY:
The prevalence of Attention Deficit/ Hyperactivity (ADHD) varies between 3 and 10% depending on the studies. Comorbidities are frequently associated, in particular anxiety disorders. School, social and family consequences of ADHD can be major, especially in the presence of a comorbidity.

The study goal is to evaluate, through questionnaires, the effect of self-hypnosis via a smartphone application, on the symptoms of inattention and anxiety in children with ADHD in addition to their treatment by methylphenidate. Parents and children complete the study questionnaires four times.

* T0: at inclusion
* T1 (T0+6 weeks): after 6 weeks of using the self-hypnosis application 5 days out of 7 for group 1 in parallel with the usual treatment / after 6 weeks of usual treatment for the group 2
* T2 (T0+8 weeks): after a wash-out period of 2 weeks (usual treatment only) for both groups
* T3 (T0+14 weeks): after 6 weeks of use of the self-hypnosis application 5 days out of 7 for group 2 in parallel with the usual treatment / after 8 weeks of usual treatment for the group 1, following the 6 weeks of use of the application.

DETAILED DESCRIPTION:
The prevalence of Attention Deficit/ Hyperactivity (ADHD) varies between 3 and 10% depending on the studies. Comorbidities are frequently associated, in particular anxiety disorders. School, social and family consequences of ADHD can be major especially in the presence of a comorbidity.

The management of ADHD requires an effective multimodal approach to attention disorders and comorbid disorders. In France, the Haute Autorité de Santé recommends the combination of drug treatment with methylphenidate (as a second line or, for serious cases, from the first line) and a non-drug treatment such as behavioral therapies, cognitive remediation and psycho-educational support.

As part of this project, and more generally for the care of young ADHD patients, it is interesting to target a method that can be deployed in a relatively controlled way in addition to other non-drug measures and without contradicting them. Hypnosis is a technique that is already widely used in the treatment of pain. In the field of mental health, the clinical use of hypnosis is a relevant strategy to support self-regulation capacities in anxious children. Indeed, this technique offers an easily accessible experience of reducing arousal and dissociating internal physical sensations and perceptions, while promoting attentional focus towards the examination of new possibilities. The repeated use of self-hypnosis incorporating imaginary exposure facilitates the feeling of capacity for action ("empowerment") in the face of anxiety-provoking elements, reduces hyper-reactivity, and leads to the control of physiological reactivity.

In France, it is difficult for families to find structures for the care and monitoring of child's ADHD. The lack of speech therapists, the waiting list in public medical institution, the cost of follow-up by private psychologists, the lack of specialized structures are obstacles to care and increase the risk of pejorative evolution. In this context, the use at home by the child of a digitized self-hypnosis tool has all its interest.

The objectives of the study are to evaluate, through questionnaires, the effect of self-hypnosis via a smartphone application, on the symptoms of inattention and anxiety in children with ADHD in addition to taking classical pharmacological load by methylphenidate.

Parents and children complete the study questionnaires four times.

* T0: at inclusion
* T1 (T0+6 weeks): after 6 weeks of using the self-hypnosis application 5 days out of 7 for group 1 in parallel with the usual treatment / after 6 weeks of usual treatment for the group 2
* T2 (T0+8 weeks): after a wash-out period of 2 weeks (usual treatment only) for both groups
* T3 (T0+14 weeks): after 6 weeks of use of the self-hypnosis application 5 days out of 7 for group 2 in parallel with the usual treatment / after 8 weeks of usual treatment for the group 1, following the 6 weeks of use of the application.

ELIGIBILITY:
Inclusion Criteria:

* Patient of French mother tongue, aged 7 to 12 with a diagnosis of ADHD made by a child psychiatrist or neuropediatrician according to DSM-5 criteria
* Patient treated with methylphenidate and followed by the child psychiatry department - Reference Center for Language and Learning Disorders of the Necker Enfants Malades Hospital
* Information and consent of holders of parental authority and of the patient

Exclusion Criteria:

* Presence of an intellectual disability
* Presence of an autism spectrum disorder

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 49 (Actual)
Dates: Start 2023-09-04 (Actual); Primary Completion 2024-06-23 (Actual); Study Completion 2024-06-23 (Actual)

PRIMARY OUTCOMES:
Change in severity of attention deficit | Day 0, 6 weeks, 8 weeks, 14 weeks
  The severity of attention deficit is assessed with the Conners 3 questionnary. It provide information's for information for 11 scales and includes 110 questions. Our research will focus on the T-score of inattention scale (mean=100, standard deviation=10). The higher the score is, the severed the symptom is. The change of the inattention scale T-score from base line at 6 weeks and 14 weeks will be used as primary outcome.

SECONDARY OUTCOMES:
Change in severity of anxiety with a self-questionnaire | Day 0, 6 weeks, 8 weeks, 14 weeks
  Assessment with the Revised-Children's Manifest Anxiety Scale (R-CMAS). The R-CMAS is a self-questionnaire of 28 anxiety items and 9 lying items. It provides scores for Total Anxiety and 4 subscales: Physiological Anxiety, Worry/Sensitivity, Social Concerns/Concentration, Lie Scale. The notation is binary: true/false. Our research will focus on anxiety total T-score (mean at 50, standard deviation at 10). The higher the T-Score is, the severed the symptom is. The change of the anxiety total R-CMAS T-score from base line at 6 weeks and 14 weeks will be used as seondary outcome.
Change in severity of anxiety with a hetero-questionnaire | Day 0, 6 weeks, 8 weeks, 14 weeks
  Assessment with the Child Behavior Checklist inventory (CBCL). The CBCL provides information on 6 scales: Anxious/Depressed, Withdrawn/Depressed, Somatic Complaints, Social Problems, Thought Problems, Attention Problems, Rule-Breaking Behavior, and Aggressive Behavior. It includes 113 questions, noted from 0 to 2, depending on the presence of each symptom. Our research will focus on the T-score of the anxiety/Depressed scale (mean at 50, standard deviation at 10). The higher the T-Score is, the severed the symptom is. The change of the inattention scale T-score of the CBCL from base line at 6 weeks and 14 weeks will be used as seondary outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Grosmaitre, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker-Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hiltunen, S., Virta, M., Salakari, A., Antila, M., Chydenius, E., Kaski, M., … Partinen, M. (2014). Better long-term outcome for hypnotherapy than for CBT in adults with ADHD: Results of a six-month follow-up. Contemporary Hypnosis and Integrative Therapy, 30, 118-134.
- [Background] Kaiser P. Childhood anxiety and psychophysiological reactivity: hypnosis to build discrimination and self-regulation skills. Am J Clin Hypn. 2014 Apr;56(4):343-67. doi: 10.1080/00029157.2014.884487. PMID 24938076
- [Background] Landier W, Tse AM. Use of complementary and alternative medical interventions for the management of procedure-related pain, anxiety, and distress in pediatric oncology: an integrative review. J Pediatr Nurs. 2010 Dec;25(6):566-79. doi: 10.1016/j.pedn.2010.01.009. Epub 2010 Mar 12. PMID 21035021
- [Background] Richardson J, Smith JE, McCall G, Pilkington K. Hypnosis for procedure-related pain and distress in pediatric cancer patients: a systematic review of effectiveness and methodology related to hypnosis interventions. J Pain Symptom Manage. 2006 Jan;31(1):70-84. doi: 10.1016/j.jpainsymman.2005.06.010. PMID 16442484
- [Background] Virta, M., Salakari, A., Antila, M., Chydenius, E., Partinen, M., Kaski, M., & Iivanainen, M. (2010). Hypnotherapy for adults with attention deficit hyperactivity disorder: A randomized controlled study. Contemporary Hypnosis, 27, 5-18.